CLINICAL TRIAL: NCT06462157
Title: The Feasibility and Effects of Group Compassionate Mind Training for Adults Experiencing the Menopause Transition: a Preliminary Investigation
Brief Title: Group Compassionate Mind Training for Adults Experiencing the Menopause Transition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26701/001
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Menopause

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online CMT groups (Experimental): Online Compassionate Mind Training
  Interventions: Other: Compassionate Mind Training
- Control Group (No Intervention): Treatment as usual

INTERVENTIONS:
Other: Compassionate Mind Training — Participants will attend 6 x 90-minute online CMT sessions. CMT is delivered by combining taught information, exercises, and practices. It is effective, so the aim is to explore its use with menopausal women.
  Other Names: CMT
  Arms: Online CMT groups

SUMMARY:
Menopause transition occurs naturally for women aged 45-55. In addition to the hormone changes, there are often changes in other areas of life including low mood, anxiety, 'brain fog' and embarrassment. Some people may not be eligible for or want to receive hormone replacement therapy, therefore psychological treatments for menopause have been investigated. There is growing evidence for the use of Compassionate Mind Training (CMT). CMT aims to reduce feelings of self-criticism and shame which are commonly reported by adults experiencing the menopause, by helping individuals to take better care of themselves, known as self-compassion. Findings show menopausal individuals who are more self-critical may be more vulnerable to difficulties during menopause. Therefore, CMT could help manage this. CMT improves self-compassion and reduces depressive symptoms, with group formats found to be more effective than individual or self-help. A previous study of online self-help CMT for the menopause received positive feedback for the therapy and people improved in several areas including self-compassion. Clearly, there could be benefits to offering CMT as a treatment for menopause. Given that group CMT is effective in other populations and groups are more economical and practical for the NHS, this study is interested in looking at the impact of group CMT on menopause.

This study aims to find out how practical and suitable group CMT is for improving the wellbeing of adults experiencing the menopause, and what their views are on the therapy and taking part in the study. To measure the aims, we will look at the ease of recruiting people to the study, whether they are happy to be randomly allocated to receive the therapy or not, whether they stay in the study, the number of completed questionnaires and feedback from participants. It will also look at whether there have been any changes in different domains e.g. anxiety and self-compassion. This will be done through a variety of quantitative and qualitative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 40-60) who are biologically female
* Women who are experiencing symptoms of the menopause or peri-menopause; which is naturally occurring. This is identified through the STRAW criteria. Individuals have to answer Yes on at least one of the STRAW screening questions to ensure women are in the perimenopause or menopausal period.
* Substantial English verbal communication and comprehension skills
* Capacity to consent
* Confident in using video conferencing applications (MsTeams)
* Willingness to take part in a post-intervention interview about their experience.
* PHQ-9 score 5-19 (mild to moderate clinical cut offs)
* GAD-7 score 5-15 (mild to moderate clinical cut offs)

Exclusion Criteria:

* People under the age of 40
* People currently receiving any form of psychology intervention.
* Transgender females who are biologically male
* More than 5 years post menopause.
* PHQ-9 score greater or equal to 20 (severe clinical cut off)
* GAD-7 score greater or equal to 15 (severe clinical cut off)

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-10-23 (Estimated); Study Completion 2026-10-23 (Estimated)

PRIMARY OUTCOMES:
The Revised Women's Health Questionnaire | To be completed within one week before and within one week after the intervention
  Measures health-related quality of life by measuring perceptions of physical and emotional experiences of middle-aged women. All subscales are scored from yes, definitely (1) to no, not at all (4) with subscales scored with a scoring algorithm transforming each score to a 0-100 scale.
36-Item Short Form Survey | To be completed within one week before and within one week after the intervention
  Measures quality of life. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
The Menopause Representations Questionnaire (MRQ) | To be completed within one week before and within one week after the intervention
  Measure to assess beliefs about menopause. It consists of 20 items, scored either no (0), uncertain (1) or yes (2). Higher scores indicate more beliefs about the menopause.
Fears of Compassion Scale | To be completed within one week before and within one week after the intervention
  Measures fears of compassion. It has 38 items, scored either dont agree at all (0) to completely agree (4) on a Likert scale. There are three subscales, subscale items are summed, with higher scores indicating higher fears of compassion.
Patient Health Questionnaire-9 (PHQ-9) | To be completed within one week before and within one week after the intervention
  Measures severity of depression. Score from 0-27, higher scores represent higher severity of symptoms of depression.
General Anxiety Disorder-7 (GAD-7) | To be completed within one week before and within one week after the intervention
  Measures severity of anxiety. Score from 0-21, higher scores represent higher severity of symptoms of anxiety.
The forms of Self Criticising/Attaching & Self-reassuring scale (FSCRS) SELF-REASSURING SCALE (FSCR | To be completed within one week before and within one week after the intervention
  Measures self criticism and the ability to self-reassure. It is a 22-item scale with the items making up three components; inadequate self, hatred self and self-reassure. Responses are given on a 5-point likert scale (0 = not at all lime me, to 4 = extremely like me). Higher scores indicate a greater sense of inadequacy (score 0-20), self-hate (score 0-16), and self-reassurance (score 0-20).

SECONDARY OUTCOMES:
Post intervention interviews | Within 5 weeks post intervention
  Qualitative data on experiences from the group

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Spector, Principal Investigator — UCL
Locations (1):
- University College London, London, County, United Kingdom

IPD SHARING:
Plan to Share IPD: No